CLINICAL TRIAL: NCT04743960
Title: Assessing Metabolic and Sleep Consequences of Overnight Home Parenteral Nutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: ASPEN Rhoads Research Foundation (Industry)
Responsible Party: Principal Investigator, Hassan Dashti, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020P003741
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Feeding Patterns; Sleep; Glucose Intolerance; Short Bowel Syndrome
Keywords: Parenteral Nutrition; Chrononutrition; Chronobiology; Nutrition Support; Sleep; Metabolomics
MeSH Terms: conditions — Feeding Behavior; Glucose Intolerance; Short Bowel Syndrome; Hyperphagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nighttime cycled parenteral feeds followed by daytime cycled parenteral feeds (Experimental): Patients will follow nighttime feeding regimen for one week, and then advance their feeds (approximately 12 hours earlier) to daytime feeding regimen for one week.
  Interventions: Dietary Supplement: Time-of-day of parenteral nutrition provision

INTERVENTIONS:
Dietary Supplement: Time-of-day of parenteral nutrition provision — Parenteral nutrition will be provided during the nighttime followed by daytime.

SUMMARY:
The purpose of this study is to determine whether advancing the timing of home parenteral nutrition from overnight to daytime regimens leads to improved glucose profiles and sleep quality, and other changes in plasma metabolic signatures.

DETAILED DESCRIPTION:
Emerging evidence suggests that considering the time-of-day in clinical care may optimize health, partly through limiting sleep disruption and circadian misalignment. Acute sleep and circadian rhythms disturbances are associated with cardiometabolic derangements, including persistent hyperglycemia, a significant contributor to life-threatening complications. However, it is currently considered standard practice for patients on parenteral nutrition to be fed for 12-hour periods overnight. Current guidelines lack explicit guidance regarding the time-of-day when nutrition support should be administered. Thus, the overall objective of the clinical trial is to comprehensively examine a novel dimension of clinical nutrition by determining whether advancing the timing of home parenteral nutrition from overnight to daytime regimens leads to improved glucose profiles and sleep quality, and other changes in plasma metabolic signatures. The study is a 2-week controlled cross-over feeding trial where 20 short bowel syndrome patients will follow their usual overnight parenteral nutrition regimen for one week, and then advance their feeds to daytime for a second week. Patients will be assessed objectively using non-invasive, novel technologies and 'omics techniques. The investigators hypothesize that advancing the timing of home parenteral nutrition feeds to a daytime regimen is a cost-efficient, effective, and feasible nutrition timing countermeasure against metabolic derangements, fragmented sleep, and decreased quality of life. Results of this study may provide evidence-based, cost-efficient, and effective nutrition support countermeasures against hyperglycemia and sleep disruption, and could potentially modify current widespread clinical nutrition support practice.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or non-pregnant female volunteers (age 18-79)
* Short bowel syndrome diagnosis
* Able and willing to give consent and comply with study procedures
* Currently on routine home parenteral nutrition (at least 6 months)

Exclusion Criteria:

* Blind, deaf or unable to speak English
* Women who are pregnant or nursing
* Diabetes diagnosis or currently taking or intending to take any diabetes medication or medications influencing sugars including oral glucocorticoids, growth hormone, erythropoietin, or chemotherapeutic
* Current use of sleep medication and melatonin
* With skin condition that precludes wearing sensors
* Within the last year, bariatric surgery or pregnancy
* Within the last one month, acute infections or illnesses requiring medical attention, hospitalizations, Emergency Department visits, blood transfusions, blood loss, blood donations
* Major changes in diet or physical activity level in the past 3 months
* Sleep and circadian disorders (such as obstructive sleep apnea and delayed sleep phase syndrome)
* Anticipated barriers or challenges to daytime and/or overnight cycled infusions

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
Change in 24-hour average glucose from nighttime to daytime feeds | Average values from days 1 to 7 (nighttime feeds) and days 8 to 14 (daytime feeds).
  Glucose will be continuously measured using continuous glucose sensors. Blood glucose will be averaged during each of the two 1-week feeding regimens (nighttime and daytime).
Change in number of interruptions of sleep by physical movement assessed by actigraphy from nighttime to daytime feeds | Actigraphy data from days 1 to 7 (nighttime feeds) and days 8 to 14 (daytime feeds).
  Sleep will be objectively measured from actigraphy. The number of interruptions of sleep by physical movement will be calculated as 100 × the number of groups of consecutive mobile 30-s epochs/by the total number of immobile epochs. This measure will reflect sleep quality.

SECONDARY OUTCOMES:
Change in area under-the-curve of glucose from nighttime to daytime feeds | Glucose values from days 1 to 7 (nighttime feeds) and days 8 to 14 (daytime feeds) during 12-hour cycled feeds.
  Glucose will be continuously measured using continuous glucose sensors. Area under-the-curve of blood glucose during the 12-hour feeds will be calculated using the trapezoid method and adjusted for baseline glucose values. Area under-the-curve of glucose will be averaged for each of the two 1-week feeding regimens (nighttime and daytime).
Change in average daily duration of glucose levels above 140 mg/dl from nighttime to daytime feeds | Average values from days 1 to 7 (nighttime feeds) and days 8 to 14 (daytime feeds).
  Glucose will be continuously measured using continuous glucose sensors. Duration of glucose levels above 140 mg/dl will be averaged during each of the two 1-week feeding regimens (nighttime and daytime).
Change in fasting insulin concentration from nighttime to daytime feeds | Blood draw scheduled on days 8 and 15.
  Serum insulin will be measured from fasting blood samples collected on day 8 and 15.
Change in sleep duration from nighttime to daytime feeds | Average values from days 1 to 7 (nighttime feeds) and days 8 to 14 (daytime feeds).
  Sleep duration will be objectively measured from actigraphy and sleep logs. Duration will be averaged will be averaged during each of the two 1-week feeding regimens (nighttime and daytime).
Change in sleep midpoint from nighttime to daytime feeds | Average values from days 1 to 7 (nighttime feeds) and days 8 to 14 (daytime feeds).
  Sleep midpoint will be objectively measured from actigraphy and sleep logs. Midpoint will be averaged will be averaged during each of the two 1-week feeding regimens (nighttime and daytime).
Change in midpoint of least-active 5h timing from nighttime to daytime feeds | Average values from days 1 to 7 (nighttime feeds) and days 8 to 14 (daytime feeds).
  Measure of sleep timing as determined from actigraphy. Timing will be averaged will be averaged during each of the two 1-week feeding regimens (nighttime and daytime).
Change in midpoint of most-active 10h timing from nighttime to daytime feeds | Average values from days 1 to 7 (nighttime feeds) and days 8 to 14 (daytime feeds).
  Measure of sleep timing as determined from actigraphy. Timing will be averaged will be averaged during each of the two 1-week feeding regimens (nighttime and daytime).

CONTACTS AND LOCATIONS:
Overall Officials: Hassan S Dashti, Ph.D., R.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dashti HS, Leong A, Mogensen KM, Annambhotla M, Li P, Deng H, Carey AN, Burns DL, Winkler MF, Compher C, Saxena R. Glycemic and sleep effects of daytime compared with those of overnight infusions of home parenteral nutrition in adults with short bowel syndrome: A quasi-experimental pilot trial. Am J Clin Nutr. 2024 Feb;119(2):569-577. doi: 10.1016/j.ajcnut.2023.11.016. Epub 2023 Dec 1. PMID 38043867
- [Background] Rahmoune A, Winkler MF, Saxena R, Compher C, Dashti HS. Comparison between self-reported and actigraphy-derived sleep measures in patients receiving home parenteral nutrition: Secondary analysis of observational data. Nutr Clin Pract. 2024 Apr;39(2):426-436. doi: 10.1002/ncp.11077. Epub 2023 Oct 1. PMID 37777983
- [Derived] Dashti HS, Sevilla-Gonzalez M, Mogensen KM, Winkler MF, Compher C. Plasma metabolomics changes comparing daytime to overnight infusions of home parenteral nutrition in adult patients with short bowel syndrome: Secondary analysis of a clinical trial. Clin Nutr ESPEN. 2024 Aug;62:28-32. doi: 10.1016/j.clnesp.2024.04.025. Epub 2024 May 13. PMID 38901946